CLINICAL TRIAL: NCT02288000
Title: Effect of a 15-day Memantine Treatment on Biomarkers of AD in Healthy Volunteers
Brief Title: Prediction of Cognitive Properties of Memantine for Neurodegenerative Diseases
Acronym: WP3_P002
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012_55; 2013-001671-21 (EudraCT Number)
Record Dates: First submitted 2014-11-06; First posted 2014-11-11 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Alzheimer Disease; Battery
Keywords: Alzheimer; Memantine; biomarkers; battery; cognition; imaging; neuropsychology
MeSH Terms: conditions — Alzheimer Disease | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Memantine (Active Comparator): Memantine will be administered OS as of 10 mg- capsule one per day in the morning over 15 days.
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator): The placebo will be presented as capsule comparable to memantine
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — Memantine will be administered OS as of 10 mg- capsule one per day in the morning over 15 days.
  Other Names: Memantine Arrow
  Arms: Memantine
Drug: Placebo — the placebo will be administered OS as of 10 mg- capsule one per day in the morning over 15 days.
  Arms: Placebo

SUMMARY:
The early assessment of new drugs for Alzheimer's disease remains difficult because of the lack of predictive end-point. The use of a battery including different parameters could improve this early development of new drugs. Nevertheless, the interest of such a battery should previously be validated with the yet marketed AD drugs.

DETAILED DESCRIPTION:
The aim of the present study is to test the effect of a 15-day treatment with memantine on a mixed battery associating cognitive assessment, imaging and neurophysiological tests in healthy volunteers.

This multicenter, randomized, placebo-controlled, cross-over study is double-blind controlled and is conducted in 3 centers located in France (Lille, Marseille and Toulouse).

18-30 years old, healthy volunteers, without any neurological or psychiatric impairment, will complete 2 test sessions in a randomized order: one with a 15-day treatment with memantine, the other with placebo, and will be submitted to a mixed battery during the 14th and 15th day of the treatment. The primary outcome of the study will be based on cognitive assessment, imaging parameters and neurophysiological parameters

ELIGIBILITY:
Inclusion Criteria:

* 18-30 year old male non-smoker subjects
* Subject without cognitive impairment or cognitive complaint (Moca>26, Mac Nair scale<15)
* Subject without history of brain disease (severe brain trauma, stroke, cerebral tumor,…)
* Subject without major medical or surgical history
* Subject without current chronic disease
* Subject without current cerebral disease
* Subject without vascular or metabolic risk factor
* Subject without history or current mental disease or addiction (MINI)
* Subject without lesion on MRI
* Subject without abnormal electrical activities on EEG
* Subject without use of chronic treatment or psychotropic drugs or substances
* French speaker subject and able to understand the test instructions

Exclusion Criteria:

* Subject with dementia or cognitive decline identified by Moca < 26
* Subject with vascular or metabolic risk factor
* Subject with history or current mental disease or addiction
* Subject with family history of young-onset dementia
* Subject with family history of chronic or severe neurological or mental disease (first degree relatives)
* Subject receiving a chronic treatment
* Subject with claustrophobia or contra-indication to MRI
* Subject unable to understand the test instructions

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-09-14 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Pharmacog battery | 15 days
  * cognitive tests (8 items of the Cantab battery) :
    * Motor screening
    * 4 tests for visual memory (Delayed Matching to Sample, Paired Associated Learning, Pattern Recognition Memory, Spatial Recognition Memory)
    * 1 test for executive functions (Spatial Working Memory)
    * 2 tests for attention (Reaction Time, Rapid Visual Information Processing)
    * completed by a modified ADNI battery : ADAScog
  * imaging
    * fMRI
    * PET-FDG
  * neurophysiological
    * EEG

CONTACTS AND LOCATIONS:
Overall Officials: Régis Bordet, MD, PhD, Study Chair — University Hospital, Lille
Locations (3):
- France (3):
  - CHRU de Lille/ Centre d'investigation Clinique, Lille
  - CIC Marseille, Marseille
  - CIC Toulouse, Toulouse